CLINICAL TRIAL: NCT03283631
Title: INTERCEPT: INTracerebral EGFR-vIII Chimeric Antigen Receptor Gene-Modified T CElls for PaTients With Recurrent GBM
Brief Title: Intracerebral EGFR-vIII CAR-T Cells for Recurrent GBM
Acronym: INTERCEPT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We are halting enrollment of this study.
Sponsor: Gary Archer Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Duke Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Gary Archer Ph.D., Assistant Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00083828; 5P50CA190991-03 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliosarcoma
Keywords: Malignant Glioma; INTERCEPT; Pro00083828; Adult; Chimeric Antigen Receptor; CAR T cell; EGFRvIII
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGFRvIII-CARs (Experimental): Gamma-retroviral MSGV1 139 scFv EGFRvIII CAR gene-modified T cells
  Interventions: Biological: EGFRvIII-CARs

INTERVENTIONS:
Biological: EGFRvIII-CARs — Gamma-retroviral MSGV1 139 scFv EGFRvIII CAR gene-modified T cells

SUMMARY:
The goal of this protocol is to transfer autologous peripheral blood mononuclear cells (PBMCs) transduced with genes encoding a chimeric antigen receptor (CAR) that recognizes epidermal growth factor receptor variant III (EGFRvIII) tumor-specific antigen into patients with recurrent glioblastoma (GBM) following stereotactic radiosurgery (SRS). The CAR used is targeted to a tumor-specific mutation of the epidermal growth factor receptor, EGFRvIII, which is expressed on a subset of patients. Normal PBMCs derived from patients with GBM are genetically engineered with a viral vector encoding the CAR and infused directly into the patient's tumor with the aim of mediating regression of their tumors. Despite our CAR being targeted to a tumor specific antigen, given the prior toxicity using CARs that were not targeted to tumor-specific antigens, the investigators elected to begin with very low doses of cells. Enrollment on this study was suspended in April 2020 while an amendment to reduce the anticipated number of participants was under review and approved. The decision to terminate the study was made in January, 2021 to shift toward the next iteration of a related CAR T cell trial.

DETAILED DESCRIPTION:
Patients with evidence of radiographic recurrence who expressed EGFRvIII on their original tumor diagnosis had autologous PBMCs harvested by leukapheresis. These autologous PBMCs were transduced with a retrovirus containing the sequences for the EGFRvIII CAR and sent to the Duke Radiopharmacy for radiolabeling with 111Indium (111In). Within 2-3 weeks of leukapheresis, on Day -4 to -2, patients had a BrainLab MRI to prepare for biopsy and catheter placement. On Day -1, the patient underwent standard of care (SOC) stereotactic biopsy under local anesthesia to confirm tumor recurrence. At the time of biopsy, prior to catheter insertion and administration of study drug, the presence of recurrent tumor was confirmed by histopathology. If tumor recurrence was confirmed, a catheter was placed intratumorally for delivery of EGFRvIII-CARs by Convection Enhanced Delivery (CED).

SRS will took place on Day 0 (+1 day) and 111In-labeled EGFRvIII-CARs were infused on the same day over a 6 to 6.5 hour period immediately after SRS.

On days 1 and 2 after 111In-labeled EGFRvIII-CAR infusion, whole planar imaging followed by Single-Photon Emission Computed Tomography (SPECT) Computed Tomography (CT) imaging assessed the intracerebral and systemic localization of the 111In-labeled EGFRvIII-CARs that described the distribution of EGFRvIII-CARs within the brain and systemically.

This protocol was designed to determine the maximum tolerated dose (MTD) of a novel, tumor-specific treatment with autologous EGFRvIII-CARs. The proposed starting dose was 2.5 x 10^8 of 111In-labeled cells in 3 milliliters (mL). The infusion flow rate was fixed at 0.5 mL/hr.

Enrollment on this study was suspended in April 2020 while an amendment to reduce the anticipated number of participants was under review and approved. Upon approval of this amendment, the enrollment suspension remained due to a change in access to necessary equipment for CAR manufacturing. The decision to terminate the study was made in January, 2021 to shift toward the next iteration of a related CAR T cell trial. The knowledge gained from this study experience is directing our next CAR T-cell platform and will be used to secure additional funding.

ELIGIBILITY:
Inclusion Criteria:

1. Disease progression or recurrence of a supratentorial World Health Organization (WHO) grade IV malignant glioma (GBM or gliosarcoma) based on imaging studies with measurable disease. At the time of biopsy, prior to stereotactic radiosurgery (SRS) and administration of the EGFRvIII-CARS, the presence of recurrent tumor must be confirmed by histopathological analysis.
2. Adults ≥ 18 years old.
3. Karnofsky Performance Status (KPS) score ≥ 70.
4. EGFRvIII, the target antigen, must be identified on tumor tissue by immunohistochemistry (IHC) or Polymerase Chain Reaction (PCR), i.e. EGFRvIII positive via pathology report.
5. Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,000 cells/µl, platelets ≥ 125,000 cells/µl (prior to biopsy).
6. Serum creatinine ≤ 1.5 mg/dl, serum glutamic oxaloacetic transaminase (SGOT), and bilirubin ≤ 1.5 times upper limit of normal (prior to biopsy).
7. Signed informed consent approved by the Institutional Review Board.
8. Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [IUD; only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to starting SRS.
9. Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.
10. Meet eligibility requirements for SRS: able to get MRI; the patient must have a lesion that, in the opinion of the study radiation oncologist, can safely receive SRS to the entire tumor; must not be abutting optic apparatus or brainstem and catheter tip will be at least 5mm away from the ventricle; and must be able to be secured and positioned in a stereotactic U-frame mask.

Exclusion Criteria:

1. Pregnant or breast-feeding.
2. Patients with known potentially anaphylactic allergic reactions to gadolinium-DTPA.
3. Patients who cannot undergo MRI with contrast or SPECT/CT.
4. Patients with evidence of tumor in the brainstem, cerebellum, optic apparatus, or spinal cord, radiological evidence of actively growing multifocal disease, or leptomeningeal disease.
5. Patients < 12 weeks from the end of radiation therapy, unless they have two progressive scans at least 4 weeks apart, have progression outside of the radiation field, or have histologic confirmation of progression.
6. Severe, active comorbidity, including any of the following:

   1. Unstable angina and/or congestive heart failure requiring hospitalization;
   2. Transmural myocardial infarction within the last 6 months;
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study initiation;
   4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy;
   5. Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
   6. Known autoimmune disorder, such as HIV;
   7. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy;
   8. Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
7. Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
8. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin;
9. Current, recent (within 4 weeks of the administration of this study agent), or planned participation in another experimental therapeutic drug study.
10. Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks) or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to biopsy unless patients have recovered from side effects of such therapy.
11. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5 F, 37.5 C).
12. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to CAR T Cell infusion.
13. Prior therapy targeted to EGFRvIII.
14. Prior history of brain SRS, (patients who have received external beam radiation per standard of care are allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) | 4 weeks
  MTD of EGFRvIII-CAR gene-modified T cells when administered intracerebrally by CED after SRS in patients with recurrent GBM

SECONDARY OUTCOMES:
Assessment of T Cell trafficking within the brain tumor | 2 days
  Change in volume of distribution and maximal percentage of enhanced tumor volume covered
Assessment of T cell trafficking systemically | 2 days
  Change in the volume of distribution of 111In-labeled EGFRvIII-CARs present in each body area (neck, chest, abdomen, pelvis, and extremities)
Median survival | 1 year
  The time between SRS / CAR treatment and death or last follow-up
Median progression-free survival | 1 year
  The time between SRS / CAR treatment and first failure (death or disease progression)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Landi, MD, Principal Investigator — Duke University; David Ashley, MBBS, FRACP, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/clinical-trials